CLINICAL TRIAL: NCT04320420
Title: Feasibility of an Adapted Physical Activity Program for Patients Treated With an Autologous Hematopoietic Stem Cell Transplantation
Brief Title: Feasibility of an Adapted Physical Activity Program for Patients Treated With an Autograft (APA²)
Acronym: APA²
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weprom (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WP-2019-05; 2019-A02203-54 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2020-03-20; First posted 2020-03-25 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Myeloma; Lymphoma; Autologous Transplant
Keywords: Adapted Physical Activity; Autograft; Sarcopenia
MeSH Terms: conditions — Neoplasms, Plasma Cell; Lymphoma; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): The APA program is defined in 3 stages:
  STEP 1: during the initial chemotherapy over 3 months
  * 3 supervised APA sessions/week on site:
    * two muscle strengthening sessions, stretching, flexibility in the gym
    * a cardio session (Nordic Walking: outdoors)
  * at home: exercise book if the patient wishes
  STEP 2: during hospitalization for the autograft, over 1 month:
  * 2 sessions/week supervised by an APA engineer + exercise book and encouragement of individual work
  * If the patient wishes, he can continue the exercises carried out with the APA engineer independently
  STEP 3: after the transplant
  * the first 3 months:
    * 2 supervised indoor sessions/week (muscle strengthening, stretching, flexibility),
    * 1-hour cardio session/week independently
  * the following 3 months: 1 indoor session per week + independent exercises at home and walking or cycling sessions
  Interventions: Other: Adapted Physical Activity

INTERVENTIONS:
Other: Adapted Physical Activity — The APA program is defined in 3 stages:
  STEP 1: during the initial chemotherapy over 3 months
  * 3 supervised APA sessions/week on site:
    * two muscle strengthening sessions, stretching, flexibility in the gym
    * a cardio session (Nordic Walking: outdoors)
  * at home: exercise book if the patient wishes
  STEP 2: during hospitalization for the autograft, over 1 month:
  * 2 sessions/week supervised by an APA engineer + exercise book and encouragement of individual work
  * If the patient wishes, he can continue the exercises carried out with the APA engineer independently
  STEP 3: after the transplant
  * the first 3 months:
    * 2 supervised indoor sessions/week (muscle strengthening, stretching, flexibility),
    * 1-hour cardio session/week independently
  * the following 3 months: 1 indoor session per week + independent exercises at home and walking or cycling sessions

SUMMARY:
Therapeutic intensification followed by an autograft of hematopoietic stem cells is a standard of care for young patients with myeloma from the first line and for lymphoma from the second or third line of treatment. This procedure remains toxic in the short and medium term with significant mortality and morbidity: the average mortality varies from 1.4 to 5%. The causes of death are linked to a severe infection, visceral bleeding or vital organ failure. This risk of mortality is partly correlated with sarcopenia.

Sarcopenia is defined by the reduction of muscle mass and strength. It was first described in the elderly and classified as geriatric syndrome such as dementia, falls or frailty. It varies from 5 to 13% between 60 and 70 years and between 11 and 50% beyond 80 years and is classified as primitive, that is to say related to age It can however be secondary to neoplasia. This event has been described in patients with hematologic malignancies during chemotherapy and can reach 55% of patients in the elderly. It is proportional to the intensity of the treatments. It emerges as an independent prognostic factor which is detrimental to survival in these patients. Physical exercise combined with nutritional support could reduce it.

The positive impact of adapted physical activity (APA) has been shown in numerous publications on reducing the incidence and risk of relapse for several cancers (breast, colon prostate). It is less obvious in hematology in view of studies published on APA with different physical activity programs depending on the time of the intervention or according to the type, duration and intensity.

The objective of this study is to assess the feasibility of an APA program in patients requiring an autologous hematopoietic stem cell transplant. It is expected that the program will have a protective effect on the appearance of induced sarcopenia and on the complications related to the procedure in the short and medium term regardless of the hematology center for patients receiving intensive treatment with support for autologous hematopoietic stem cells.

This is a feasibility study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years,
2. Patient with lymphoma or myeloma justifying an autograft of hematopoietic stem cells whatever the line of treatment,
3. Patient affiliated to a social security scheme,
4. Patient who has given written consent before any specific procedure related to the study

Exclusion Criteria:

1. Central and / or peripheral neurological deficit not allowing adapted physical activity sessions to be carried out,
2. Uncontrolled hypertension,
3. Left ventricular Ejection Fraction <50%,
4. Chronic respiratory insufficiency with alterations in the functional respiratory investigations,
5. Active viral infection: hepatitis B, C and HIV,
6. Pregnancy or breastfeeding,
7. Persons deprived of their liberty or under guardianship
8. Dementia, mental alteration or psychiatric pathology which could compromise the patient's informed consent and / or compliance with the protocol and follow-up of the trial,
9. Patient who can't follow protocol for psychological, social, family or geographic reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of an adapted physical activity program surrounding an autograft | 6 months post-autograft
  Proportion of patients performing all sessions offered per week and who performed exercises at home

SECONDARY OUTCOMES:
To assess the impact of an adapted physical activity program on the number of patients with sarcopenia following an autograft | 6 months post-autograft
  Number of patients with sarcopenia within 6 months of autograft
To assess quality of life | 12 months post-autograft
  Change in score of the Quality of Life Questionnaire (General, 30 questions) of European Organisation for the Research and Treatment of Cancer. All of the scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems
To assess fatigue | 12 months post-autograft
  Change in score of the multidimensional fatigue inventory questionnaire (20-100 with higher scores mean a worse outcome).
To assess sexual function | 12 months post-autograft
  Brief Index of Sexual Function for Women (5-75 with higher scores mean a better outcome).
To assess sexual function | 12 months post-autograft
  Male Sexual Health Questionnaire for men, Brief Index (5-125 with higher scores mean a better outcome).
To assess patient's satisfaction | 6 months post-autograft
  Specific questionnaire for study (6-25 with higher scores mean a better outcome).
To assess progression free survival | 28 months
  Time between the inclusion date and the date of the first exam who show the progression of the disease
To assess the response rate | 28 months
  Number of patients with a partial or complete response according to Lugano criteria for lymphoma and IMWG (International Myeloma Working Group) for myeloma
To assess the global physical activity load by patient and by session | 6 months post-autograft
  Calculated by Foster method
To assess the prevalence of endocrinal disorder | 28 months
  Number of patients with endocrinal disorder between the date of inclusion and the date of end of study at the numerator and the number of patients following at the denominator
To assess the prevalence of autograft's complication | 28 months
  Number of patients with autograft's complication at the numerator and the number of patients following at the denominator
To assess the duration and the cost of the hospitalization for the autograft | 6 months
  Hospitalizations will be quote (economic data) by medical information department of center
To assess the delay the period for resuming professional activity for the patients concerned, after the autograft | 28 months
  Delay between the date of autograft and the date of resuming professional activity

CONTACTS AND LOCATIONS:
Overall Officials: Katell LE DU, MD, Principal Investigator — Centre Jean Bernard/Clinique Victor Hugo
Locations (2):
- France (2):
  - CHU, Angers
  - Centre Jean Bernard/Clinique Victor Hugo, Le Mans

IPD SHARING:
Plan to Share IPD: No